CLINICAL TRIAL: NCT05276921
Title: Assessment of the Prognostic Value of the Thickness of the Quadriceps and Abdominal Muscles Measured by Ultrasound for 28-day Mortality in Postoperative ICU Patients
Acronym: SARCOPENIE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: DRANSART BOUDINA 2019
Record Dates: First submitted 2022-02-28; First posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-02

CONDITIONS: Sarcopenia ICU Ultrasound
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient: Postoperative ICU patient
  Interventions: Other: ultrasound

INTERVENTIONS:
Other: ultrasound — Quadriceps and abdominal muscle ultrasonography

SUMMARY:
Ultrasound measurement of muscle thickness, particularly of the quadriceps, can be used to highlight a reduction in lean mass. Sarcopenia is annvoluntary loss of lean mass, and it is a frequent and major problem in the intensive care unit (ICU). Sarcopenia is associated with significant morbidity and mortality, as previously demonstrated by CT scan measurements.

Nevertheless, due to its nature and cost, it does not appears reasonable to perform CT sarcopenia evaluation in all ICU patients. Described in the literature as evolving rapidly upon admission to ICU, accurate assessment of this loss of muscle mass would allow early detection of sarcopenia and adaptation of therapeutic management, particularly nutritional and rehabilitative.

There are many advantages to evaluating sarcopenia by ultrasound measurement: simple, rapid, achievable at the patient's bedside, no exposure to radiation, non-invasive, and low cost. The abdominal muscles (external oblique, internal oblique, transverse) constitute the accessory respiratory muscles. Easily accessible by ultrasound, they are a potential target for the evaluation of sarcopenia, which could be responsible for ventilatory withdrawal failures, prolonged stays in intensive care and associated complications. The combined ultrasound measurement of the quadriceps and accessory respiratory muscles in ICU patients therefore appears to be an innovative approach. Considering the ease of implementation, the validity of ultrasound (confirmed in the literature), and the safety of the technique, we wish to evaluate the link between the muscle mass at arrival in the postoperative Intensive Care Unit of the Dijon University Hospital by ultrasound measurement of the quadriceps and accessory respiratory muscles, and: mortality, duration of mechanical ventilation, length of stay and occurrence of intercurrent events.

ELIGIBILITY:
Inclusion Criteria:

* Person who has not opposed (or non-opposition of health care proxy for patients who are comatose or under the influence of sedative drugs) after receiving information about the study
* All adult patients admitted to the postoperative intensive care unit.

Exclusion Criteria:

* Protected adult or minor
* Pregnant or breastfeeding woman
* Lower limb amputation
* Refusal to participate of the patient or health care proxy
* Patient with pre-existing neuromuscular condition, tetra or paraplegia
* Morbid obesity as defined by BMI ≥ 40
* BPCO stage ≥ 3; heart failure with LVEF < 50%; patients with symptomatic valvulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: postoperative ICU patient
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
Ultrasound mesure of thickness of quadriceps and abdominal muscles | at inclusive

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France